CLINICAL TRIAL: NCT07068308
Title: Development and Effectiveness of a Wed-based FRAIL-SM Program Among Patients With Heart Failure
Brief Title: Effects of a Wed-based FRAIL-SM Program Among Patients With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NYCU113069AE
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: frailty; heart failure; self-management; web-based frailty self-management program; knowledge; family caregiver; quality of life
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wed-based FRAIL-SM program (Experimental): Patients in the intervention group will receive an 8-week web-based FRAIL-SM program including family involvement, self-regulation, autonomy support, information sharing and linkage.
  Interventions: Behavioral: web-based FRAIL-SM program
- control group (No Intervention): Patients in this group will receive usual care.

INTERVENTIONS:
Behavioral: web-based FRAIL-SM program — The 8-week web-based FRAIL-SM includes family involvement, self-regulation, autonomy support, information sharing and linkage.
  Arms: wed-based FRAIL-SM program

SUMMARY:
This study aims to examine the effects of web-based FRAIL-SM (Family involvement, self-Regulation skills training, Autonomy, Information sharing and Linkage, Self-Management) on frailty, self-management behaviors and quality of life in patients with heart failure and their families' heart failure knowledge, confidence, strain, and quality of life. Patients are recruited with a convenience sampling from two medical centers in Taiwan. The web-based FRAIL-SM includes Family involvement, self-Regulation, Autonomy support, Information sharing and Linkage.

DETAILED DESCRIPTION:
A randomized controlled trial is conducted. Subjects are selected using a convenience sampling and are randomly assigned to the intervention or control group by stratified randomization according to participation of post-acute care. Patients in the intervention group will receive an 8-week web-based FRAIL-SM program. Data is collected by researchers using a structural questionnaire including frailty, heart failure knowledge, self-care of heart failure, and quality of life and physical indicators such as levels of B-type natriuretic peptide, hemoglobin, hematocrit, albumin at baseline, 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment.

ELIGIBILITY:
Patients criteria:

Inclusion Criteria:

1. Aged above 20.
2. Diagnosed with heart failure or LVEF<40%.
3. Clear consciousness, can communicate with Chinese and Taiwanese.
4. Consent to join in this study and have family partner.
5. Access to computer or smartphone
6. Meet one of the Study of Osteoporotic Fractures of frailty

Exclusion Criteria:

1. Bed-ridden or unable to perform activities of daily living independently.
2. Diagnosed with cognitive, psychiatric disease, or major depression.
3. Acute disease condition e.g. infection or thrombosis.
4. Contraindications of performing exercise such as uncontrolled hypertension, uncontrolled arrhythmia.
5. severe neurodegenerative or muscular diseases, e.g. parkinson's disease, arthritis.

Family criteria:

Inclusion criteria

1. Aged above 20.
2. Clear consciousness, can communicate with Chinese and Taiwanese.
3. Consent to join in this study and willing to accompany with patients.
4. Access to computer or smartphone

Exclusion Criteria:

1. Bed-ridden or unable to perform activities of daily living independently.
2. Diagnosed with cognitive, psychiatric disease, or major depression.
3. Have employment relationship with patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Frailty Assessment Scale for Heart Failure scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline Frailty Assessment Scale for Heart Failure scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Frailty Assessment Scale for Heart Failure contains 15 items, each item use Likert scale four point scoring (0-3), the total scores ranged from 0 to 45, the higher scores indicate higher levels of frailty.
Changes in Dutch Heart Failure Knowledge Scale scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline Dutch Heart Failure Knowledge Scale scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Dutch Heart Failure Knowledge Scale contains 15 items. The total scores ranged from 0 to 15, the higher scores indicate higher levels of knowledge.
Changes in Self-Care of Heart Failure Index scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline Self-Care of Heart Failure Index scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Self-Care of Heart Failure Index contains 22 items, three subscales: self-care maintenance, self-care management, self-care confidence. Each subscale scores ranged from 0 to 100, the higher scores indicate higher levels of self-care maintenance, self-care management, self-care confidence.
Changes in Minnesota Living with Heart Failure questionnaire scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline Minnesota Living with Heart Failure questionnaire scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Minnesota Living with Heart Failure questionnaire contains 21 items, each item scores ranged from 0 to 5. The total socre ranged from 0 to 105, the higher scores indicate higher levels of impact on quality of life.

SECONDARY OUTCOMES:
Changes in World Health Organization Quality of Life - BREF (WHOQOL-BREF) scale scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline World Health Organization Quality of Life - BREF (WHOQOL-BREF) Scale scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The WHOQOL-BREF scale contains 28 items, four dimensions. Each dimension scores ranged from 4 to 20, the higher scores indicate higher levels of quality of life.
Changes in Caregiver Strain Index scores | baseline, 4 weeks, 8 weeks, 12 weeks and 24 weeks
  Changes from baseline Caregiver Strain Index scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Scale contains 13 items, the total scores ranged from 0 to 13, the higher scores indicate higher levels of strain.

OTHER OUTCOMES:
Changes in Hospital Anxiety and Depression Scale scores | baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Changes from baseline Hospital Anxiety and Depression Scale scores to at 4 weeks, 8 weeks, 12 weeks and 24 weeks after enrollment. The Hospital Anxiety and Depression Scale contains 14 items, two subscales: anxiety and depression. Each subscale scores ranged from 0 to 21, the higher scores indicate higher levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No